CLINICAL TRIAL: NCT00979199
Title: Evaluation of Integrated Cardiac Imaging for the Detection and Characterization of Ischemic Heart Disease
Brief Title: Evaluation of Integrated Cardiac Imaging in Ischemic Heart Disease
Acronym: EVINCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Danilo Neglia, MD, Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EVINCI; European Commission (Other Grant/Funding Number: European Commission, FPVII Health Grant N. 222915); FPVII grant 222915
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Ischemic Heart Disease
Keywords: IHD; CAD; Non invasive imaging; SPECT; PET; CMR; Echocardiography
MeSH Terms: conditions — Myocardial Ischemia

ARMS (1):
- Non invasive cardiac imaging (Other): Intervention: Non invasive cardiac imaging. 'Anatomical' information provided by CTCA is obtained in every patient together with the 'functional' information provided by stress radionuclide cardiac imaging (SPECT or PET), to assess myocardial perfusion, and/or by stress MRI or ECHO imaging to assess myocardial contraction.
  Interventions: Other: Non invasive cardiac imaging

INTERVENTIONS:
Other: Non invasive cardiac imaging — Non invasive cardiac imaging consists of CTCA combined with one Stress Imaging Test

SUMMARY:
Main purpose of the study:

To comparatively assess the diagnostic performance of non invasive anatomical and functional imaging modalities to detect significant obstructive coronary artery disease as demonstrated at invasive coronary angiography and functional evaluation of coronary lesions (fractional flow reserve).

DETAILED DESCRIPTION:
Objectives of the study

1. To test the accuracy of anatomical and functional non-invasive cardiac imaging in the diagnosis of IHD. To this purpose the "anatomical" information provided by CTA is obtained in every patient together with the "functional" information provided by stress radionuclide cardiac imaging (SPECT or PET), to assess myocardial perfusion, and/or by stress MRI or ECHO imaging to assess myocardial contraction. Non-invasive results are tested against invasive reference standards. The latter consists of invasive coronary angiography integrated by invasive measurement of fractional flow reserve (to assess the hemodynamic relevance of intermediate coronary stenoses).
2. To test the accuracy of integrated models, including clinical variables, risk factors and circulating biomarkers, to predict significant obstructive coronary artery disease in patients with chronic angina-like symptoms. To correlate biohumoral profiles with the coronary anatomical-functional phenotype as obtained by non invasive imaging in the same patients. To reach these goals the clinical characterization of patients (collected before non-invasive imaging) and the laboratory characterization (that includes novel biomarkers of cardiovascular risk) are compared with patient characterization derived from non invasive "anatomic-functional" imaging and with invasive diagnosis of significantly obstructive coronary disease.
3. To develop an advanced clinical and imaging reporting tool in cardiology. An informatics platform is developed to synthetically and clearly present the integrated clinical and imaging diagnostic profile of individual patients. A multimodal imaging reporting tool is developed including tools for "image fusion" of different imaging modalities (CT, SPECT, PET, MRI).
4. To define the most cost-effective work-up for the diagnosis and characterization of IHD. To this purpose the costs and the procedural risks (including radiation exposure) of non-invasive and invasive diagnostic procedures are prospectively collected. Cost-benefit and cost-effectiveness analyses is conducted alongside the EVINCI-study clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intermediate (>20%, <90%) risk of IHD based on age,gender,symptoms and exercise stress test results

Exclusion Criteria:

* Age < 30 Yrs or > 75 yrs
* Pregnancy (suspected or ascertained)
* LV Dysfunction (LVEF < 35% by Echo or other method)
* Low (< =20%) or high (>=90%) probability of CAD
* Acute Coronary Syndrome
* Prolonged (> 20 minutes) chest pain
* De novo or accelerated angina
* Hemodynamic or electrical instability
* Recent ST-T segment or T wave changes of ischemic nature
* Acute myocardial infarction with or without ST segment elevation
* Elevated serum cardiac markers of necrosis
* Known diagnosis of CAD
* Previously known myocardial infarction
* Previous PCI
* Previous CABG
* Persistent atrial fibrillation or advanced AV Block
* Asthma or chronic treatment with aminophylline
* Recent (<6 months) cerebral ischemic attack
* Known significant carotid stenosis or vascular aneurisms
* Asthma or chronic treatment with aminophylline
* Active cancer
* Severe hypertension. Patients cannot withdraw therapy for 12 hours.
* Congenital heart disease
* Significant valvular disease
* Cardiomyopathy (e.g. DCM, HCM, ARVC, Amyloidosis)
* Inability to provide an informed consent

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 697 (Actual)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danilo Neglia, MD, PhD, Principal Investigator — Fondazione Toscana G. Monasterio, Pisa, Italy
Locations (16):
- U.Turku, Turku, Finland
- APHP, Paris, France
- Germany (2):
  - KAE Goeppingen, Göppingen
  - TUM, Munich
- Italy (5):
  - Ospedale Versilia, Viareggio, Lucca
  - UniGE, Genova
  - UniNA, Naples
  - CNR, Pisa
  - FGM, Pisa
- LUMC, Leiden, Netherlands
- NIC, Warsaw, Poland
- Spain (2):
  - Huvhebron, Barcelona
  - SERMAS, Madrid
- UZH, Zurich, Switzerland
- United Kingdom (2):
  - QUEEN MARY Hospital London, London
  - RBHT, London

REFERENCES:
- [Derived] Caselli C, De Caterina R, Smit JM, Campolo J, El Mahdiui M, Ragusa R, Clemente A, Sampietro T, Clerico A, Liga R, Pelosi G, Rocchiccioli S, Parodi O, Scholte A, Knuuti J, Neglia D; EVINCI and SMARTool. Triglycerides and low HDL cholesterol predict coronary heart disease risk in patients with stable angina. Sci Rep. 2021 Oct 20;11(1):20714. doi: 10.1038/s41598-021-00020-3. PMID 34671067
- [Derived] Caselli C, Del Turco S, Ragusa R, Lorenzoni V, De Graaf M, Basta G, Scholte A, De Caterina R, Neglia D. Association of PCSK9 plasma levels with metabolic patterns and coronary atherosclerosis in patients with stable angina. Cardiovasc Diabetol. 2019 Oct 31;18(1):144. doi: 10.1186/s12933-019-0949-3. PMID 31672148
- [Derived] Carpeggiani C, Picano E, Brambilla M, Michelassi C, Knuuti J, Kauffman P, Underwood SR, Neglia D; EVINCI Study Investigators. Variability of radiation doses of cardiac diagnostic imaging tests: the RADIO-EVINCI study (RADIationdOse subproject of the EVINCI study). BMC Cardiovasc Disord. 2017 Feb 16;17(1):63. doi: 10.1186/s12872-017-0474-9. PMID 28202051
- [Derived] Neglia D, Rovai D, Caselli C, Pietila M, Teresinska A, Aguade-Bruix S, Pizzi MN, Todiere G, Gimelli A, Schroeder S, Drosch T, Poddighe R, Casolo G, Anagnostopoulos C, Pugliese F, Rouzet F, Le Guludec D, Cappelli F, Valente S, Gensini GF, Zawaideh C, Capitanio S, Sambuceti G, Marsico F, Perrone Filardi P, Fernandez-Golfin C, Rincon LM, Graner FP, de Graaf MA, Fiechter M, Stehli J, Gaemperli O, Reyes E, Nkomo S, Maki M, Lorenzoni V, Turchetti G, Carpeggiani C, Marinelli M, Puzzuoli S, Mangione M, Marcheschi P, Mariani F, Giannessi D, Nekolla S, Lombardi M, Sicari R, Scholte AJ, Zamorano JL, Kaufmann PA, Underwood SR, Knuuti J; EVINCI Study Investigators. Detection of significant coronary artery disease by noninvasive anatomical and functional imaging. Circ Cardiovasc Imaging. 2015 Mar;8(3):e002179. doi: 10.1161/CIRCIMAGING.114.002179. PMID 25711274

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CTCA and PET or SPECT and ECHO or MRI
Started | 697
Completed | 475
Not Completed | 222

BASELINE CHARACTERISTICS:
Arm/Group | CTCA and PET or SPECT and ECHO or MRI
Number analyzed (Participants) | 475
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9)
Sex/Gender, Customized [Number; unit: participants]
  Male | 291
  Female | 184
Region of Enrollment [Number; unit: participants]
  France | 28
  Finland | 71
  Poland | 36
  Spain | 61
  Germany | 35
  United Kingdom | 27
  Switzerland | 67
  Italy | 150

OUTCOME MEASURES:

1. Primary Outcome: Diagnosis of IHD at Invasive Coronary Angiography and FFR Measurement
Description: The outcome measure is the number of participants who received the diagnosis of IHD at invasive coronary angiography coupled with FFR measurements (in case of intermediate coronary lesions).
Time Frame: 3 months from enrollment
Measure: Number; unit: participants
Groups:
- Non Invasive Cardiac Imaging: All patients are submitted to non invasive cardiac imaging. 'Anatomical' information provided by CTA is obtained in every patient together with the 'functional' information provided by stress radionuclide cardiac imaging (SPECT or PET), to assess myocardial perfusion, and/or by stress MRI or ECHO imaging to assess myocardial contraction. All patients with at least one positive functional test undergo invasive coronary angiography to obtain the final diagnosis of IHD (Outcome measurement).
Arm/Group | Non Invasive Cardiac Imaging
Number analyzed (Participants) | 475
participants | 140

2. Secondary Outcome: Cost-benefit and Cost-effectiveness Analysis
Description: Different non invasive imaging modalities are compared in terms of a cost-effectiveness analysis where costs include direct and indirect costs incurred as a consequence of the use of each modality or combination of modalities and effectiveness is the diagnostic accuracy with invasive diagnosis of IHD as end-point.
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Non Invasive Cardiac Imaging
Serious Adverse Events (participants affected / at risk) | 0/475
Other Adverse Events (participants affected / at risk) | 5/475
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non Invasive Cardiac Imaging (N=475)
Severe chest pain (Cardiac disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No